CLINICAL TRIAL: NCT03353974
Title: The Role of Video Games Therapy on Balance and Cognitive Functions in Mild to Moderate Impaired Multiple Sclerosis Patients. A Pilot Randomized Controlled Trial.
Brief Title: Video Games Therapy on Balance and Cognitive Functions in Mild to Moderate Impaired Multiple Sclerosis Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Sofia Straudi, MD, University Hospital of Ferrara
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MS_Video_Games_Therapy
Record Dates: First submitted 2017-11-16; First posted 2017-11-27 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Video game therapy; Balance; Cognitive functions; Dual tasking
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video game therapy (Experimental): Subjects belonging to the experimental group will receive a Video Game Therapy (VGT) protocol using the Xbox console. They will receive 12 sessions of treatment within 4 weeks (3 sessions per week); each session will last 1 hour. To manage possible absence lasting one or more treatment sessions, a potential window of 5 weeks will be set to ensure the achievement of all 12 sessions. Will be required to concentrate in games whose major purposes are increasing balance, selective attention and attention shifting. During sessions the patient will be carefully controlled by a researcher who will prevent the risk of falling
  Interventions: Device: Video game therapy
- Balance platform therapy (Active Comparator): Subjects belonging to the control group will receive the same amount of therapy (12 sessions) using a balance platform (Biodex Medical Systems, Inc., Shirley, NY). Balance/rebalancing, postural stability and weight-shifting exercises ill be administered with and without visual feedback. During the first session, the tasks will be performed at an "entry level," and the exercise progression will be adjusted over time according to the patients' functional level (intermediate and difficult level). Balance platform therapy offered visual feedback and knowledge of performance (augmented feedback). The physiotherapist, as during VGT, provided additional external feedback.
  Interventions: Device: Balance platform therapy

INTERVENTIONS:
Device: Video game therapy — Video game therapy will be delivered with a commercial video game console (X-Box 360 Kinect, Microsoft, Inc., Redmond, WA).
  Arms: Video game therapy
Device: Balance platform therapy — Balance/rebalancing, postural stability and weight-shifting exercises with and without visual feedback will be administered using a balance platform (Biodex Medical Systems, Inc., Shirley, NY).
  Arms: Balance platform therapy

SUMMARY:
Multiple Sclerosis (MS) is often characterized by the presence of balance and cognitive impairments. Cognitive functions play a key role in balance control. Simultaneously performing cognitive tasks decreases walking and balance ability (Dual-Task cost). Rehabilitative treatment of patients with MS does not have to consider separately the motor and cognitive aspects. Video-Game Therapy (VGT) is a novel tool that allows a multimodal training approach. VGT typically provides augmented feedback during training that can contribute to learning motor skills. The main objective of this exploratory study will be to test the effects of a commercially available VGT on balance and cognitive function in ambulatory MS patients compared to a standardized balance platform training (BPT). Secondary, we will explore the effects of VGT and BPT on other domains that are usually impaired in MS population and that can be improved by motor rehabilitation, such as psychological well-being, fatigue and Quality of Life.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of MS (primary or secondary progressive, relapsing-remitting), without relapses in the preceding 3 months
* mild to moderate balance impairments with increased fall risk, defined as TUG > 8.4s
* disability rate definited by Kurtzke Expanded Disability Status Scale (EDSS) score from 4 to 5.5,

Exclusion Criteria:

* other conditions that may affect motor function
* impaired cognitive functioning (Mini Mental Status Examination score less than 24)
* visual impairments (daltonism and visual acuity deficit)
* medical conditions that might interfere with the ability to complete the study protocol safely.

A group of healthy subjects matched for age and sex will be involved for a comparison on the instrumental data (force platforms).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Timed Up and Go (TUG) test | Changes from baseline to end of treatment (4 weeks), following changes after 12 weeks follow up
  TUG measures balance and functional mobility.

SECONDARY OUTCOMES:
Four Square Step Test (FSST) | Changes from baseline to end of treatment (4 weeks), following changes after 12 weeks follow up
  The FSST is a timed test, intended to challenge the rapid change in direction while stepping forward, backward and sideways over a low obstacle.
Functional Reach Test (FRT) | Changes from baseline to end of treatment (4 weeks), following changes after 12 weeks follow up
  The FRT assesses the subject's stability by measuring the maximum distance an individual can reach forward while standing in a fixed position.
Dynamic Gait Index (DGI) | Changes from baseline to end of treatment (4 weeks), following changes after 12 weeks follow up
  Clinical tool to assess gait, balance and risk of fall.
Modified Fatigue Impact Scale (MFIS) | Changes from baseline to end of treatment (4 weeks), following changes after 12 weeks follow up
  Questionnaire which evaluates the perceived impact of fatigue on the subscales physical, cognitive and psychosocial functioning.
Multiple Sclerosis Walking Scale-12 (MSWS-12) | Changes from baseline to end of treatment (4 weeks), following changes after 12 weeks follow up
  This questionnaire assesses the impact of MS on walking ability.
Multiple Sclerosis Impact Scale-29 (MSIS-29) | Changes from baseline to end of treatment (4 weeks), following changes after 12 weeks follow up
  This is an health-rated quality of life questionnaire that assesses the impact of MS on physical and psychological functions.
Beck Depression Inventory-Second Edition (BDI-II) | Changes from baseline to end of treatment (4 weeks), following changes after 12 weeks follow up
  This is a 21-item self-report instrument that serves to assess depression severity
State Trait Anxiety Inventory (STAI-Y) | Changes from baseline to end of treatment (4 weeks), following changes after 12 weeks follow up
  STAI-Y is an easy-to-use and interpretative tool to detect and measure anxiety.
Go-No Go - Test of Attentional Performance T.A.P. | Changes from baseline to end of treatment (4 weeks), following changes after 12 weeks follow up
  Go-No Go task examine the specific capacity to suppress an inadequate reaction.
Test of Attentional Performance T.A.P. | Changes from baseline to end of treatment (4 weeks), following changes after 12 weeks follow up
  In this task divided attention can be explored with computerized "dual-task" test where two stimuli (visual and acoustic) are required simultaneously
Stroop Color-Word Test (SCWT) | Changes from baseline to end of treatment (4 weeks), following changes after 12 weeks follow up
  The SCWT explores sustained attention and some aspects of executive function.
Symbol Digit Modalities Test (SDMT) | Changes from baseline to end of treatment (4 weeks), following changes after 12 weeks follow up
  The SDMT consists of orally substituting a number for a pseudorandom sequence of geometric figures as quickly as possible for testing executive functions.
Instrumented Basic Balance Evaluation (IBBE) | Changes from baseline to end of treatment (4 weeks), following changes after 12 weeks follow up
  Force platform measurement are used as objective markers of subjects' balance ability.
Instrumented Dual Task (IDT) | Changes from baseline to end of treatment (4 weeks), following changes after 12 weeks follow up
  Dual cognitive-motor tasks are often used in clinical practice to evaluate the interaction between patients' cognitive and motor ability .

CONTACTS AND LOCATIONS:
Overall Officials: Sofia Straudi, MD, PhD, Study Director — Ferrara Rehabilitation Hospital
Locations (2):
- Italy (2):
  - Sofia Straudi, Ferrara, Emilia-Romagna
  - Ferrara University Hospital, Ferrara

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baroni A, Fregna G, Milani G, Severini G, Zani G, Basaglia N, Straudi S. Video game therapy on mobility and dual tasking in multiple sclerosis: study protocol for a randomised controlled trial. BMJ Open. 2021 Oct 21;11(10):e052005. doi: 10.1136/bmjopen-2021-052005. PMID 34675018